CLINICAL TRIAL: NCT06600035
Title: Gastric Ultrasound in Elective Surgical Diabetic Patients
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR801/8/24
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastric Ultrasound; Elective Surgery; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I - Diabetic: Diabetic patients
  Interventions: Device: Gastric ultrasound
- Group II - Non-diabetic: Non-diabetic patients
  Interventions: Device: Gastric ultrasound

INTERVENTIONS:
Device: Gastric ultrasound — A curved array, low-frequency (2-5 MHz) transducer providing a scan depth up to 30 cm will be used. Patients will be scanned in the supine position followed by right lateral decubitus (RLD) position. The sonographic appearance of the gastric antrum will be classified as Grade 0,1 or 2, signifying empty antrum, fluid detected in RLD position only and antral fluid in both supine and RLD positions, respectively, based on the appearance in both the positions. Cross-sectional area (CSA) will be calculated by using two perpendicular diameters-anteroposterior (AP) and craniocaudal (CC) and the formula for area of an ellipse:CSA = (AP × CC × π)/4

SUMMARY:
The aim of this study is to evaluate the role of gastric ultrasound in elective surgical diabetic patients.

DETAILED DESCRIPTION:
Aspiration of gastric contents during perioperative period is a grave complication with significant morbidity and mortality. The overall incidence of gastric content aspiration ranges between <0.1% and 19% and aspiration pneumonia account for 9% of all anesthesia-related mortality. Mendelson described the pathophysiological mechanisms of pulmonary aspiration, which led to the development of strategies to prevent pulmonary aspiration.

Consequently, American Society of Anesthesiologists (ASA) released preoperative fasting guidelines for healthy patients undergoing elective surgery, in order to reduce gastric content volume and minimize the risk of aspiration. However, there are still many situations where the ASA fasting guidelines may be not suitable, including urgent or emergency situations and medical conditions such as diabetes mellitus.

Ultrasound is widely available and has been proven to be a reliable, bedside assessment tool for real-time evaluation of gastric contents. As diabetic patients are prone to have an inadequately empty stomach even after an adequate fasting, ultrasound can be used prior to induction for screening the fasting gastric volume (GV) of diabetic patients and see if it is more than the recommended safe limit.

As a novel point-of-care application, ultrasound sonography allows anesthesiologists to evaluate a patient's gastric content and volume at the bedside and helps guide anesthetic and airway management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Undergoing elective surgery.

Exclusion Criteria:

* American Society of Anesthesiology (ASA) physical status >III.
* Body mass index (BMI) outside the range of 18.5-40 Kg/m2.
* History of upper gastrointestinal disease or previous surgery on the esophagus, stomach, or upper abdomen.
* Abnormalities of the upper gastrointestinal tract, such as gastric tumors and recent upper gastrointestinal bleeding (within the preceding 1 month).
* Taking preoperative medicines that may delay gastric emptying (e.g., anticholinergic agents, opioids).
* Hypothyroidism.
* Current smoking history.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This case-control study will be carried out on 130 cases, aged ≥ 18 years, undergoing elective surgery at Tanta University Hospitals after approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Antral cross-sectional area (CSA) | Just before surgery
  Cross-sectional area (CSA) will be calculated by using two perpendicular diameters-anteroposterior (AP) and craniocaudal (CC) and the formula for area of an ellipse:
  CSA = (AP × CC × π)/4

SECONDARY OUTCOMES:
Gastric volume | Just before surgery
  The gastric volume will be calculated using the previously validated formula:
  GVe (gastric volume in ml) = 27.0 + [14.6 × right - lateral CSA (cm2)] - (1.28 × age)
Gastric volume/weight | Just before surgery
  Gastric volume/weight will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author